CLINICAL TRIAL: NCT00216489
Title: A Non Interventional Post Authorization Safety Study (PASS) On The Rabeprazole's Administration To Adults With Gastro-Oesophageal Reflux Disease (GORD)
Brief Title: A Study of the Safety of Rabeprazole Administered to Adults With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Cilag Pharmaceutica S.A.C.I., Greece (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003502
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux; Heartburn
Keywords: gastroesophageal reflux; heartburn; rabeprazole; GERD; anti-ulcer agents; proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Rabeprazole

INTERVENTIONS:
Drug: rabeprazole sodium

SUMMARY:
The purpose of the study is to confirm the safety and effectiveness of rabeprazole in the treatment of patients with erosive or ulcerative gastroesophageal reflux disease (GERD) in routine primary health care.

DETAILED DESCRIPTION:
Gastroesophageal reflux can result in mild to severe symptoms in some persons. Heartburn, a burning sensation or discomfort rising behind the breastbone, is a common symptom. Gastroesophageal reflux disease (GERD) can be described as a condition with clearly identified clinical symptoms or the change in tissue structure that results from the reflux of contents from the stomach or small intestine into the esophagus. This is a study to confirm the safety and effectiveness of rabeprazole in the treatment of patients with GERD in routine primary health care. The study has two phases. Patients will receive treatment with rabeprazole tablets once daily for 8 weeks. In the second phase, patients will be monitored by their physician for a follow up period to end of study (12 months). Safety assessments include the incidence of adverse events throughout the treatment and follow up phases, and physical examination and laboratory tests at end of treatment and after 4 months. Assessments of effectiveness include the degree of relief of symptoms at beginning and end of treatment and at specific intervals during follow up. The study hypothesis is that rabeprazole is well-tolerated with long term treatment of patients with GERD in routine primary health care. Rabeprazole tablet (20 milligrams[mg]) once daily in the morning for 8 weeks. Dose may be increased to 2 tablets daily (40 mg maximum) at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of erosive or ulcerative gastroesophageal reflux disease (GERD) during at least a period of 3 months prior to study initiation and symptoms of GERD for at least 3 days per week within the 2 weeks prior to study initiation. The symptoms of erosive or ulcerative gastroesophageal reflux disease includes the following: heartburn, aching behind the breastbone, a need for antacids, and difficulty in swallowing. Patients with evidence by endoscopy of erosive or ulcerative gastroesophageal reflux disease with no Barret-type tissue transformation.

Exclusion Criteria:

* No narrowing or inflammation of the esophagus
* no known gastro-duodenal ulcer
* no infections (other than H. Pylori), inflammations or hemorrhage of the stomach, small or large intestine
* no prior surgery of the stomach or intestine
* no known history of primary kinetic disorders of the esophagus, other than GERD
* no history of enlarged veins of the esophagus or stomach
* no pregnant or nursing females, or those lacking adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2003-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events throughout treatment (8 weeks) and follow up (12 months)

SECONDARY OUTCOMES:
Severity of symptoms at baseline and specified intervals during treatment and follow up, rated from "no problem" to "very severe problem"; physical examination and laboratory tests at end of treatment and after 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pharmaceutica S.A.C.I. Clinical Trial, Study Director — Janssen-Cilag Pharmaceutica S.A.C.I.